CLINICAL TRIAL: NCT04133506
Title: Defining a PGE2 Pathway in Regulating Eczema
Brief Title: PGE2/IL-22 Pathway in Various Forms of Eczema
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 19/SS/0094
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema | interventions — Aspirin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- acute eczema: acute eczema patients with eczema <72 hours no drugs
- chronic eczema: chronic eczema with eczema > 72 hours no drugs
- allergic contact dermatitis: allergic contact dermatitis with a clear allergen identified no drugs
- psoriasis patients: patients with plaque psoriasis no drugs
- healthy volunteers: dithranol or DNCB (used to induce irritant or allergic eczema used safely in similar research studies for decades) aspirin to half the group to assess the effects on downstream mediators
  Interventions: Drug: Aspirin 300mg

INTERVENTIONS:
Drug: Aspirin 300mg — see earlier (only half of healthy volunteers receive aspirin)
  Groups: healthy volunteers

SUMMARY:
Objectives: Eczema is a chronic inflammatory skin condition characterised immunologically by T cellmediated inflammation. The pathogenic mechanisms involved in its development are incompletely understood and targeted treatment options are limited. The investigators will study the Prostaglandin E2 (PGE2)/IL22/IL17 pathway which plays an important role in murine model chronic skin inflammation. The investigators wish to identify subtypes of human eczema in which this pathway may be involved and to determine whether manipulation of this pathway may offer effective new treatments.

Design, tissue/cells, techniques and measurements: To address these objectives, the investigators will measure the expression of IL22, IL17A and PGE2 synthases and receptors in skin biopsies from eczema and psoriasis patients using immunohistochemistry (confirming this with RT-PCR). IL22/IL17 producing Tcells (from peripheral blood) and their skin-homing capability (by ex-vivo cell culture and flow cytometry) will be measured. Deriving immune cells from skin biopsies using Villanova's technique1, the investigators will determine the T-cell response to PGE2 looking at PGE2 receptors and cytokine expression, interrogating these cells by flow cytometry. To determine the sequence and kinetics of activation of the PGE2/IL22/IL17 pathway the investigators will measure each immune mediator at specific time points by recruiting healthy volunteers inducing irritant and allergic contact dermatitis using dithranol and DNCB respectively. The investigators will repeat the experiment dividing volunteers into two arms, one pre-treated for one week with a non-specific prostaglandin inhibitor (aspirin) and the second with a placebo control.

DETAILED DESCRIPTION:
Defining a specific IL-22-mediated pathway in regulating eczema (i) Introduction: Overarching aim: Eczema is a significant chronic skin disease yet the need for targeted treatments remains largely unmet. In this study, I will investigate the cellular mechanisms for how the IL-22 pathway contributes to skin inflammation in eczema and whether pharmacologic manipulation of this pathway might offer effective new treatments for this common disease.

Main hypothesis and objectives: I hypothesise that prostaglandin E2 (PGE2) promotes eczema through activating IL-22 signalling and that blockade of PGE2 receptors EP2/EP4 reduces eczema severity. I will interrogate this hypothesis with three objectives: (1) to examine whether IL22 overexpression in eczema patients is driven by endogenous PGE2 acting via EP2 and EP4 receptors, (2) to determine whether this PGE2-IL-22 pathway is of particular importance in distinct subtypes of eczema and, (3) to study whether blocking EP2/EP4 receptors upstream of IL-22 and IL-17 will reduce eczema severity.

Background and importance of research:

Eczema is the most common chronic inflammatory skin disease, with a rising prevalence in Western society placing an increasing economic burden on the health service.3 It is increasingly being recognised as a heterogenous disease encompassing acute and chronic eczema, and allergic contact dermatitis (ACD). It cumulatively affects over 4% of adults and 10% of children of whom 50% have persistent disease in adulthood. The recent UK Translational Research Network in Dermatology priority setting exercise highlighted the burden created by this common and important disease.The requirement for a greater understanding of eczema pathogenesis according to subtype allowing patient stratification, and the dearth of treatment options available are significant unmet needs. This is in contrast with advances made in the development of biological therapies for psoriasis although refinement of these was also prioritised.

Atopic eczema may predispose children to the "atopic march", and early effective treatment may reduce progression to asthma and hayfever in these patients. Understanding the immune pathway in eczema may provide insight into inflammatory pathways generic to a range of diseases especially those arising at the environmental allergen/epithelial interface.

The mainstay of treatment for eczema over the last 50 years has been topical corticosteroids and latterly calcineurin inhibitors with the particular side effects of, respectively, skin thinning and carcinogenesis.

Topical treatments are useful in mild disease but lack efficacy in those with moderate or severe eczema. Systemic immunosuppressants are used for moderate and severe disease, but these are 'blunderbuss' drugs, with no specificity for eczema and as a result can cause an extensive range of potentially serious adverse effects. Dupilumab, the first biologic treatment targeting dysregulated elements of the immune system in eczema has just received its European Marketing Authorisation approval. The trial data are impressive and confirm that immune-targeting eczema treatments will, produce a genuine paradigm shift in treatment of this disabling disease, yet 30% of patients do not respond. This highlights the importance of an increased understanding of immune dysfunction in eczema and the finding of new potentially 'druggable' targets.

Th22 cells are the predominant inflammatory infiltrative cells in chronic eczema lesional skin, and IL-22 produced by Th22 and Th17 cells induces pathognomonic epidermal hyperplasia and also reduction of filaggrin expression, leading to epithelial barrier disruption in a self-amplifying loop.

Th22 infiltration correlates directly with eczema severity, and IL22 gene expression is increased in atopic dermatitis, suggesting IL-22 inhibition therapies as a specific target for eczema. It is believed that IL-22 is as important a 'driver' cytokine in eczema as IL-17 has been in psoriasis.

Confirmation of the importance of IL-22 in driving eczema has been the phase 2a clinical trial showing successful treatment of severe eczema with an anti-lL-22 antibody (fezakinumab).

Chronic eczema and psoriasis share some immunological features. In particular, IL-17 and IL-22 are upregulated in both, although IL-17 predominates in psoriasis while IL-22 predominates in chronic eczema. Specific IL-17 antagonists are highly effective treatments for psoriasis but not eczema. Both cytokines may be upregulated by PGE2, but shared pathways of induction are not fully understood.

Therefore, identification of molecules or pathways that specifically regulate IL-22/IL-17 signaling will be particularly valuable because these approaches might offer new therapeutic strategies for treating eczema and also psoriasis.

As a well-known inflammatory mediator, PGE2, is one such molecule. The investigators have published data from a completely separate from this study (i.e. not results from this study), the investigators have previously shown that PGE2, through its receptors EP2 and EP4, promotes IL-22/IL-17 production from both innate and adaptive lymphocytes and mediates chronic inflammation in numerous tissues including skin. The investigators have shown that by either pharmacologically inhibiting endogenous PGE2 production with a COX inhibitor, indomethacin, or by genetically blocking EP4 signaling, hapten (oxazolone, OXA)-induced chronic allergic contact dermatitis in mice is reduced, and this is correlated with reduction of IL-22+CD4+ cells in skin-draining lymph nodes. The phenotype of the imiquimod mouse model resembles eczema and psoriasis.

PGE2/IL23 (as it impacts on IL-17 and IL-22) represents an elegant therapeutic target for both eczema and psoriasis in mice (imiquimod mouse model) with similar potential in man. In a study which is completely separate to this (not results of this study) it was shown (published data) that genes related to IL-22/IL-17 and PGE2 signaling pathways are up-regulated in close correlation in inflammatory skin in both eczema and psoriasis.

ELIGIBILITY:
Inclusion Criteria:

-

Eczema patients must meet criteria of one of the following groups:

Have eczema and attend the Edinburgh Dermatology Clinic.

The normal control patients will be matched for age and sex as closely as possible to our eczema patients.

The participants should be able to give informed consent and should be at least 16 years of age with no upper limit.

Psoriasis patients:

The participants will have a diagnosis of psoriasis and attend Edinburgh Dermatology clinic.

Controls will be age and gender matched. There is no upper age limit, but the lower age limit is 16.

Healthy volunteers:

The participants should have no intolerance or allergy to aspirin and no allergy/sensitivity to dithranol or DNCB.

There is no upper age limit but the lower age limit is 16.

Exclusion Criteria:

-

Eczema patients:

1. Treatment with systemic corticosteroids or other immune response modifying systemic drugs such as azathioprine or methotrexate 2 months before the study starts.
2. Inability to give informed consent.

Psoriasis:

1. Treatment with systemic corticosteroids or other immune response modifying systemic drugs such as azathioprine or methotrexate 2 months before the study starts.
2. Inability to give informed consent.

For healthy volunteers:

1. intolerance/allergy to aspirin and allergy/sensitivity to dithranol or DNCB.
2. involvement in another study at the same time.
3. pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will require 12 from each of the three eczema groups: acute, chronic and Allergic Contact Dermatitis as well as 4 psoriasis patients and 4 samples from plastic surgery patients. This comes to a total of 44 patients.
  For healthy controls undertaking the dithranol/DNCB study the investigators will anticipate a group of 8 and when the investigators repeat the experiment and administer aspirin the investigators will divide these 8 patients into 4 who receive aspirin (a non-selective prostaglandin inhibitor) and 4 who do not receive aspirin.
  44 patients (including the banked healthy skin of plastic surgery patients) +8 healthy volunteers= 52 as above.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Laboratory assessment of skin and blood of patients | 3 years
  We wish to determine if PGE2 and IL22 levels in skin and blood are elevated in specific subtypes of eczema by measuring this in their skin and blood when not receiving any treatments. This will take the form of measuring protein levels of PGE2 and IL-22 in blood and skin. This will allow us to stratify patients according to those in whom PGE2 and IL-22 is over-expressed (we don't expect this to be elevated in all patients) and will enable us to determine who we could treat in clinical trial in the future with future therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Weller, MB BCh, Principal Investigator — NHS and University of Edinburgh
Locations (1):
- QMRI, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
only if ethically permissible and unquestionably relevant to the eczema community and for patient benefit